CLINICAL TRIAL: NCT06756022
Title: Prospective, Multicenter, Real-world Study of Dolasetron Mesylate Injection for the Prevention of Chemotherapy-induced Nausea and Vomiting in Children With Acute Lymphoblastic Leukemia
Brief Title: Dolasetron for the Prevention of CINV in Children With Acute Lymphoblastic Leukemia
Status: Recruiting | Type: Observational
Sponsor: Anhui Provincial Children's Hospital (Other)
Responsible Party: Principal Investigator, Tianping Chen, Associate chief physician, Anhui Provincial Children's Hospital
Other Study IDs: EYLL-2024-036
Record Dates: First submitted 2024-12-21; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Chemotherapy Induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — dolasetron

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Use of dolasetron mesylate injection to prevent nausea and vomiting induced by chemotherapy: Subjects with childhood acute lymphoblastic leukemia treated with dolasetron mesylate injection for the prevention of nausea and vomiting induced by induction chemotherapy
  Interventions: Drug: Dolasetron mesylate injection

INTERVENTIONS:
Drug: Dolasetron mesylate injection — 1.8 mg/kg Dolasetron mesylate injection should be injected intravenously 30±10 min before chemotherapy infusion, with the maximum dose not exceeding 100 mg. It can also be mixed with apple juice or apple-grape juice for oral use, the oral dose is 1.8 mg/kg, the maximum amount is not more than 100 mg, taken orally within 1 h before chemotherapy.
  Other antiemetic drugs, except dolasetron, are at the discretion of the subject's supervising physician in accordance with clinical practice.

SUMMARY:
This is a prospective, multicenter, real-world study of 500 participants with childhood acute lymphoblastic leukemia who are scheduled to receive dolasetron mesylate injection for prophylaxis against chemotherapy-induced nausea and vomiting.

This study did not make any decision or process intervention for clinical antitumor therapy. The study plans to observe the control of nausea and vomiting within 120 h (D1-D5) after receiving induction chemotherapy and the safety within 7 days (or until this discharge, whichever occurs first).

During the whole study, demographic data, history of motion sickness, ECOG score, complications, name and dosage of anti-tumor therapy drugs, this antiemetic regimen, nausea and vomiting, rescue therapy drugs, combined drugs and adverse events were recorded.

DETAILED DESCRIPTION:
Screening period: D-14~D0 (D1 recorded on the day of chemotherapy drug infusion)

Subjects who planned to receive induction chemotherapy for the first time signed informed consent for this study, completed screening period examination, checked the inclusion criteria before drug infusion, and successfully screened subjects received CINV（chemotherapy-induced nausea and vomiting） prophylaxis regimen including Dolasetron mesylate injection.

Treatment observation period: D1~D5 (beginning of study drug administration - 120 h after chemotherapy drug infusion)

Subjects who met all inclusion criteria and did not meet any exclusion criteria were required to complete pre-chemotherapy CINV prophylaxis 30±10 min before induction chemotherapy drug infusion, as described in the administration protocol. The time of starting infusion of chemotherapy drugs (referring to other chemotherapy drugs except hormone drugs in the chemotherapy regimen) was recorded as 0 h, and the subsequent days were calculated as 24 hours.

Within 120 h after the start of chemotherapy infusion, if the subject had at least one episode of vomiting, retching, or nausea and complained of antiemetic therapy, the investigator evaluated the subject and gave remedial antiemetic therapy, which was determined by the investigator.

Within 120 h after the infusion of chemotherapy drugs, the subject or guardian will fill in the occurrence of vomiting/retching and nausea daily through the subject's diary. If there were any omissions in the subjects' diaries, the researchers would remind the subjects to fill in the contents through phone calls and wechat.

Follow-up period: D6~D7 (or until this discharge, whichever occurs first)

Adverse events were collected from D6 to D7 after chemotherapy drug infusion began (or until this discharge, whichever occurred first), and the relevant data were recorded in the study medical records and EDC（Electronic Data Capture） system.

ELIGIBILITY:
Inclusion Criteria:

1. Age 2~17 years old
2. The diagnosis of acute lymphoblastic leukemia was analyzed by comprehensive examination of bone marrow cell morphology, immune typing, cytogenetics and molecular biology.
3. The subjects plan to receive induced remission therapy such as VDLP/VDLD+CAM, multicenter CCCG ALL 2015 protocol, SCCCG-ALL-2023 protocol, etc. according to Guidelines for Diagnosis and Treatment of Childhood acute lymphoblastic Leukemia (2018 Edition) for the first time
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score 0-2
5. Expected to survive for more than 3 months
6. Subject or guardian can read, understand and complete subject diary.

Exclusion Criteria:

1. Allergic to Dolasetron mesylate injection and its excipients
2. Patients with prolonged QTc interval (QT interval ≥460 ms)
3. Other conditions considered by the researchers not to be included in the group.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Nausea and vomiting induced by induction chemotherapy in children with acute lymphoblastic leukemia
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Response (CR) rate during 0-120 hour after chemotherapy (global phase) | 0-120 hour after chemotherapy
  CR defined as no vomiting or retching occurring within 120 hours after chemotherapy and no remedial medication being used

SECONDARY OUTCOMES:
Response (CR) rate 0-24 hour after chemotherapy (acute phase) | 0-24 hour after chemotherapy
  CR defined as no vomiting or retching occurring within 24 hours after chemotherapy and no remedial medication being used
Response (CR) rate 24-120 hour (delayed period) after chemotherapy | 24-120 hour after chemotherapy
  CR defined as no vomiting or retching occurring within 24-120 hours after chemotherapy and no remedial medication being used
Proportion of subjects who did not vomit at 0-24 hour and 24-120 hour after chemotherapy | 0-24 hour and 24-120 hour after chemotherapy
  Data were derived from subjects' diaries；Vomiting defined as even when very small amounts of stomach contents are expelled or retching （muscle movements in which vomiting occurs but stomach contents are not expelled)
Proportion of subjects who did not use rescue treatment 0-24 hour and 24-120 hour after chemotherapy | 0-24 hour and 24-120 hour after chemotherapy
  Data were derived from subjects' diaries；Rescue treatment includes commonly used antiemetic drugs, decided by the investigator
0-120 h after chemotherapy when vomiting (vomiting or retching) first occurs or rescue treatment is given (whichever occurs first) | 0-120 hour after chemotherapy
  Data were derived from subjects' diaries；Vomiting defined as even when very small amounts of stomach contents are expelled or retching （muscle movements in which vomiting occurs but stomach contents are not expelled)；Rescue treatment includes commonly used antiemetic drugs, decided by the investigator
Proportion of subjects free of nausea 0-24 hour and 24-120 hour after chemotherapy | 0-24 hour and 24-120 hour after chemotherapy
  Data were derived from subjects' diaries
The incidence and severity of adverse events (aes) within 7 days after chemotherapy (or until this discharge, whichever occurs first) | 7 days after chemotherapy (or until this discharge, whichever occurs first)
  Adverse reactions were judged by the investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Children's Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No